CLINICAL TRIAL: NCT04671498
Title: Detection by Circulating RNA With Optimized Machine Learning Technology for Breast Cancer: DROPLET-BC Study
Brief Title: Droplet-BC Screening Test for the Detection of Breast Cancer, the DROPLET-BC Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Preferred Medicine, Inc (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0724; NCI-2020-08583 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0724 (Other: M D Anderson Cancer Center); MOD00009113 / IC-1243721 (Other: Roswell Park Comprehensive Cancer Center)
Record Dates: First submitted 2020-12-04; First posted 2020-12-17 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ancillary-correlative (biospecimen collection) (Breast Cancer patients): Participants undergo collection of blood sample for the Droplet-BC test. All participants' medical records are also reviewed.
  Interventions: Procedure: Biospecimen Collection; Procedure: Droplet-BC Test; Other: Electronic Health Record Review
- Ancillary-correlative (biospecimen collection) (Volunteer): Participants undergo collection of blood sample for the Droplet-BC test. All participants' medical records are also reviewed.
  Interventions: Procedure: Biospecimen Collection; Procedure: Droplet-BC Test; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood sample
Procedure: Droplet-BC Test — Undergo Droplet-BC Test
Other: Electronic Health Record Review — Medical records are reviewed

SUMMARY:
This study investigates if a new type of test called Droplet-BC screening test can classify breast cancer patients from non-cancer volunteers by circulating small-noncoding RNA in the blood with a statistical validity. This study also investigates if this test can classify the subgroup of breast cancer patients with a variety of conditions. Information from this study may provide a new method of breast cancer screening/diagnosis

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the sensitivity and specificity of the Droplet-BC screening test for distinguishing breast cancer (BC) patients from non-cancer volunteers, using reference data confirmed at sites.

SECONDARY OBJECTIVES:

I. To determine the performance (sensitivity and specificity) of the Droplet-BC screening test for the classification of early-stage BC.

II. To determine the performance (sensitivity and specificity) of the Droplet-BC screening test for classifying patients into non-cancer volunteer (Breast Imaging-Reporting and Data System [BI-RADS] Categories 1 and 2) and BC patient subgroups.

III. To determine the performance (sensitivity and specificity) of the Droplet-BC screening test to classify different subgroups between non-cancer volunteers (BI-RADS category 1) versus BC patients plus non-cancer volunteers (BI- RADS category 2).

IV. To determine the performance (sensitivity and specificity) of the Droplet-BC screening test for the classification of non-cancer volunteers into BI-RADS categories 0-5 (small cohort study).

V. To determine the performance (sensitivity and specificity) of the Droplet-BC screening test for the multi-classification among cancer stage.

VI. To compare the sensitivity of the Droplet-BC test with mammogram for detecting BC by extracting a subgroup of BC patients that have mammogram results.

VII. To compare the sensitivity of the Droplet-BC test with ultrasound for detecting BC by extracting a subgroup of BC patients that have ultrasound results.

VIII. To compare the sensitivity of the Droplet-BC test with MRI for detecting BC by extracting a subgroup of BC patients that have magnetic resonance imaging (MRI) results.

IX. To conduct all analyses described above with subgroups of participants matched as closely as possible for age, race/ethnicity, cancer history, current medication, family history of cancer, and/or breast cancer gene (BRCA) status.

EXPLORATORY OBJECTIVES:

I. To evaluate the sensitivity and specificity of the Droplet-BC test to detect cancer among different age groups.

II. To evaluate the sensitivity and specificity of the Droplet-BC test to detect cancer among individuals of differing ethnicities.

III. To compare expression levels of small ribonucleic acid (RNAs) among different age groups.

IV. To compare expression levels of small RNAs among individuals of differing ethnicities.

OUTLINE:

Participants undergo collection of blood sample for the Droplet-BC test. Breast cancer patients' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* BREAST CANCER PATIENTS: Newly diagnosed with breast cancer
* BREAST CANCER PATIENTS: Not received cancer treatment for newly diagnosed with breast cancer
* BREAST CANCER PATIENTS: Able to comprehend, sign, and date the written informed consent document to participate in the study
* BREAST CANCER PATIENTS: Able and willing to provide a one-time blood sample
* BREAST CANCER PATIENTS: Age >= 18 years old
* NON-CANCER VOLUNTEERS: Have undergone a screening mammogram
* NON-CANCER VOLUNTEERS: Not currently taking any drugs for cancer treatment or any cancer prevention medication
* NON-CANCER VOLUNTEERS: Able to comprehend, sign, and date the written informed consent document to participate in this study
* NON-CANCER VOLUNTEERS: Able and willing to provide blood samples according to provided written instructions
* NON-CANCER VOLUNTEERS: Seen by a provider (physician or advanced practice nurse [APN]) in the Cancer Prevention clinic at MD Anderson Cancer Center or other participating sites
* NON-CANCER VOLUNTEERS: Age >= 18 years old

Exclusion Criteria:

* BREAST CANCER PATIENTS: Known current pregnancy
* BREAST CANCER PATIENTS: History of breast cancer treatment in the past
* BREAST CANCER PATIENTS: Participation in any interventional clinical study within the previous 30 days in which an experimental treatment is administered or might be administered through a randomized assignment of the subject to one or more study groups
* BREAST CANCER PATIENTS: Any condition that, in the opinion of the investigator, should preclude participation in the study
* NON-CANCER VOLUNTEERS: Known current pregnancy
* NON-CANCER VOLUNTEERS: History of breast cancer (breast ductal carcinoma in situ [DCIS] and invasive)
* NON-CANCER VOLUNTEERS: History of any cancer except non-melanoma skin cancer and cervical dysplasia
* NON-CANCER VOLUNTEERS: Participation in any interventional clinical study within the previous 30 days in which experimental treatment is administered or might be administered through a randomized assignment of the subject to one or more study groups
* NON-CANCER VOLUNTEERS: Any condition that in the opinion of the investigator, should preclude participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients and non-cancer volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the Droplet-BC screening test for detecting breast cancer | Up to study completion (estimated 18 months)
  Assessed within subgroups of participants determined by cancer history, medication, family history of cancer, and/or BRCA status.
Specificity of the Droplet-BC screening test for detecting breast cancer | Up to study completion (estimated 18 months)
  Assessed within subgroups of participants determined by cancer history, medication, family history of cancer, and/or BRCA status.

SECONDARY OUTCOMES:
Sensitivity of the Droplet-BC screening test for the classification of early-stage breast cancer (BC) | Up to study completion (estimated 18 months)
  Early-stage means breast ductal carcinoma in situ (DCIS) stage and stage I/II BC. Assessed within subgroups of participants determined by cancer history, medication, family history of cancer, and/or BRCA status.
Specificity of the Droplet-BC screening test for the classification of early-stage breast cancer | Up to study completion (estimated 18 months)
  Early-stage means DCIS stage and stage I/II BC. Assessed within subgroups of participants determined by cancer history, medication, family history of cancer, and/or BRCA status.
Sensitivity of the Droplet-BC screening test for the classification of patients into non-cancer volunteer (Breast Imaging Reporting and Data System [BI-RADS] categories 1 and 2) and BC patient subgroups | Up to study completion (estimated 18 months)
  Assessed within subgroups of participants determined by cancer history, medication, family history of cancer, and/or BRCA status.
Specificity of the Droplet-BC screening test for the classification of patients into non-cancer volunteer (BI-RADS categories 1 and 2) and BC patient subgroups | Up to study completion (estimated 18 months)
  Assessed within subgroups of participants determined by cancer history, medication, family history of cancer, and/or BRCA status.
Sensitivity of the Droplet-BC screening test for the classification of different subgroups between non-cancer volunteers (BIRADS category 1) and BC patients plus non-cancer volunteers (BI-RADS category 2) | Up to study completion (estimated 18 months)
  Assessed within subgroups of participants determined by cancer history, medication, family history of cancer, and/or BRCA status.
Specificity of the Droplet-BC screening test for the classification of different subgroups between non-cancer volunteers (BIRADS category 1) and BC patients plus non-cancer volunteers (BI-RADS category 2) | Up to study completion (estimated 18 months)
  Assessed within subgroups of participants determined by cancer history, medication, family history of cancer, and/or BRCA status.
Sensitivity of the Droplet-BC screening test for the classification of non-cancer volunteers into BI-RADS categories 0-5 (small cohort study) | Up to study completion (estimated 18 months)
  Assessed within subgroups of participants determined by cancer history, medication, family history of cancer, and/or BRCA status.
Specificity of the Droplet-BC screening test for the classification of non-cancer volunteers into BI-RADS categories 0-5 (small cohort study) | Up to study completion (estimated 18 months)
  Assessed within subgroups of participants determined by cancer history, medication, family history of cancer, and/or BRCA status.
Sensitivity of the Droplet-BC screening test for the classification of BC patients into cancer stages 0-IV | Up to study completion (estimated 18 months)
  Assessed within subgroups of participants determined by cancer history, medication, family history of cancer, and/or BRCA status.
Specificity of the Droplet-BC screening test for the classification of BC patients into cancer stages 0-IV | Up to study completion (estimated 18 months)
  Assessed within subgroups of participants determined by cancer history, medication, family history of cancer, and/or BRCA status.
Sensitivity of the Droplet-BC test compared with mammogram for detecting BC by extracting a subgroup of BC patients that have mammogram results | Up to study completion (estimated 18 months)
  Assessed within subgroups of participants determined by cancer history, medication, family history of cancer, and/or BRCA status.
Sensitivity of the Droplet-BC test compared with ultrasound for detecting BC by extracting a subgroup of BC patients that have ultrasound results | Up to study completion (estimated 18 months)
  Assessed within subgroups of participants determined by cancer history, medication, family history of cancer, and/or BRCA status.
Sensitivity of Droplet-BC test compared with magnetic resonance imaging (MRI) for detecting BC by extracting a subgroup of BC patients that have MRI results | Up to study completion (estimated 18 months)
  Assessed within subgroups of participants determined by cancer history, medication, family history of cancer, and/or BRCA status.

CONTACTS AND LOCATIONS:
Overall Officials: Naoto T Ueno, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org